CLINICAL TRIAL: NCT06268119
Title: Effectiveness of Postoperative Delirium Prevention, Diagnosis and Intervention Protocol on Patients Monitored in the Intensive Care Unit After Cardiac Surgery
Brief Title: Effectiveness of Delirium Care Protocol After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonul Kara Soylemez (Other)
Responsible Party: Sponsor-Investigator, Gonul Kara Soylemez, Instructor, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MustafaKU-SBF-GKS-01
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Delirium, Postoperative
Keywords: delirium; cardiac surgery; nursing
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: The control group received standard care. The intervention group received care in line with postoperative delirium prevention, diagnosis, and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standard clinical care) (No Intervention): Control group receiving standard care administered by doctors and nurses for delirium management in the intensive care unit
- Intervention group (care with protocol) (Experimental): The intervention group received care in line with the postoperative delirium prevention, diagnosis and intervention protocol after the delirium training given by the researcher to intensive care unit nurses.
  Interventions: Other: training nurses and caring for patients to prevent, diagnose, and intervene in postoperative delirium.

INTERVENTIONS:
Other: training nurses and caring for patients to prevent, diagnose, and intervene in postoperative delirium. — The intervention group received care in line with the postoperative delirium prevention, diagnosis and intervention protocol after the delirium training given by the researcher to intensive care unit nurses.
  Arms: Intervention group (care with protocol)

SUMMARY:
This study was conducted as a quasi-experimental study to determine the effectiveness of the postoperative delirium prevention, diagnosis and intervention protocol in patients monitored in the intensive care unit after cardiac surgery.

DETAILED DESCRIPTION:
This study was conducted as a quasi-experimental study to determine the effectiveness of the postoperative delirium prevention, diagnosis and intervention protocol in patients monitored in the intensive care unit after cardiac surgery. The research was conducted at Antalya Training and Research Hospital between 06.03.2023 and 22.05.2023. The sample of the study consisted of 64 patients who underwent cardiac surgery and met the inclusion criteria. Within the scope of the study, patients were divided into two groups: control (32) and intervention (32). While the patients in the intervention group received care in line with the "Postoperative delirium prevention, diagnosis and intervention protocol", the patients in the control group received routine nursing care for delirium. The data of the study were collected using the Patient Identification Form, Acute Physiological and Chronic Health Evaluation, Glasgow Coma Scale, Richmond Agitation-Sedation Scale, Confusion Assessment Scale in the Intensive Care Unit, Nurse Diagnosis Form, Information Assessment Form for Postoperative Delirium (Pretest-Posttest) and Postoperative Delirium Prevention, Diagnosis and Intervention Protocol Checklist. In the first stage of the study, which consisted of three stages, the incidence of delirium in the control group patients receiving routine nursing care and the delirium diagnosis status of the nurses were determined. In the second stage, nurses were given training on postoperative delirium prevention, diagnosis and intervention protocol, and a preliminary study of the protocol was conducted. In the third phase, which is the last phase, patients in the intervention group received care in line with the "Postoperative Delirium Prevention, Diagnosis and Intervention Protocol".

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being 18 years or older,
* Ability to speak and communicate in Turkish,
* Having undergone cardiac surgery and being on the first postoperative day,
* Richmond Agitation and Sedation Scale (RASS) score of -3 and above,
* Having a Glasgow Coma Scale (GCS) score of 8 and above,
* Not having a serious psychiatric or neurological diagnosis,
* No serious visual or auditory problems

Exclusion Criteria:

* Undergoing surgeries other than cardiac surgery (such as abdominal endovascular aneurysm repair, thoracic endovascular aneurysm repair, deep vein thrombosis, peripheral artery disease, carotid endarterectomy),
* Previous cardiac surgery,
* Postponing or canceling the surgery,
* No preoperative admission to the cardiovascular surgery service and no emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Scale in the Intensive Care Unit (CAM-ICU) | Three weeks
  With the application of CAM-ICU, an evaluation is made as "there is delirium" or "there is no delirium". CAM-ICU; It consists of four items including sudden change of consciousness or fluctuation in the patient's level of consciousness, attention assessment, and evaluation of thought organization and level of consciousness. According to this scale, in order for patients to be diagnosed with delirium, the first and second items and one of the third or fourth items must result in favor of delirium.

SECONDARY OUTCOMES:
Glasgow Coma Scale (GCS) | Three weeks
  It is used to evaluate the patients' state of consciousness. With a scale consisting of three parts: eye opening, motor and verbal response, the patients' response to stimuli in these three areas is evaluated and scored. It is evaluated between three and fifteen points, with fifteen points indicating full consciousness and three points indicating deep coma. In order for CAM-ICU to be applied to patients, the GCS score must be eight or above. If the GCS score is eight or below, the patient is considered to be in a coma and cannot be evaluated.
Richmond Agitation-Sedation Scale (RASS) | Three weeks
  Before starting the delirium evaluation, the state of consciousness (alertness) is first evaluated. RASS takes values between "(+4)" and "(-5)". While the ideal level where the patient is alert and calm is scored as "0" on the scale, positive RASS scores "(+1,+2,+3,+4)" indicate an agitated patient; Negative RASS scores "(-1,-2,-3,-4,-5)" indicate patients who are sedated or in a coma.
Information Assessment Form for Postoperative Delirium (Pretest-Posttest) | One week
  The knowledge assessment form for postoperative delirium (Pretest-Posttest) was developed by researchers by scanning the literature in order to measure the knowledge levels of nurses working in intensive care units before and after training on postoperative delirium. For each item in the form consisting of 30 questions, answers were received from the participants as "True", "False" and "I don't know". "1" point was given for each "True" statement, and "0" point was given for each "False" and "I don't know" statements. The highest score that can be obtained from the test is "30". The form, consisting of items regarding the definition of delirium, risk factors, symptoms, prevention, diagnosis and intervention of delirium, was applied by the researcher to all nurses who attended the training before and after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Kara Soylemez, MD, Principal Investigator — Mustafa Kemal University
Locations (1):
- Antalya Training and Research Hospital, Antalya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Allen SR, Frankel HL. Postoperative complications: delirium. Surg Clin North Am. 2012 Apr;92(2):409-31, x. doi: 10.1016/j.suc.2012.01.012. PMID 22414419
- [Background] Hshieh TT, Inouye SK, Oh ES. Delirium in the Elderly. Clin Geriatr Med. 2020 May;36(2):183-199. doi: 10.1016/j.cger.2019.11.001. PMID 32222295
- [Derived] Soylemez GK, Bulut H. The effectiveness of postoperative delirium prevention, diagnosis, and intervention protocol in patients monitored in the intensive care unit after cardiac surgery: a quasi-experimental study. BMC Nurs. 2024 Dec 18;23(1):904. doi: 10.1186/s12912-024-02547-y. PMID 39695628